CLINICAL TRIAL: NCT02014324
Title: Complete Endosonographic Staging of Lung Cancer: a Systematic Single Scope Approach
Brief Title: Single Scope Staging of Lung Cancer With Endosonography
Acronym: SCORE
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL42787.018.13
Record Dates: First submitted 2013-05-30; First posted 2013-12-18 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Indication Mediastinal Staging; Complete Endosonography
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- (suspected) NSCLC, mediastinal staging, endosonography: Patients with potentially medically operable and resectable NSCLC are eligible if there is an indication for pathological evaluation of mediastinal lymph nodes.
  Interventions: Procedure: Endosonography

INTERVENTIONS:
Procedure: Endosonography — Complete endosonographic mediastinal staging is performed in 2 steps:
  1. Systematic EBUS (airways)
  2. Systematic EUS-B (esophagus)
  Other Names: EBUS; EUS-B

SUMMARY:
Rationale: Lung cancer is the most commonly diagnosed cancer worldwide and is the most frequent cause of cancer death. Accurate staging is important because it directs treatment and prognosis. Mediastinal staging can be done by both EBUS-TBNA and EUS-FNA. These two techniques have a complementary diagnostic range and the combined procedure is suited for assessment of almost the entire mediastinum. In practice, when mediastinal tissue staging is indicated, endoscopists often perform either an EBUS or an EUS investigation (instead of the combined procedure). Second, frequently only one or two, by imaging suspected lymph node stations, are sampled (ie. targeted approach).

Objectives: main and secondary:

1. Complete endosonographic (combined endobronchial and esophageal) staging using a single EBUS scope improves locoregional staging (N2, N3, T4) versus EBUS staging alone.
2. Systematic mediastinal staging results in improved locoregional staging compared to PET-CT directed assessment of the mediastinum (ie targeted approach).

Study population: Patients with potentially operable and resectable NSCLC are eligible if there is an indication for mediastinal nodal sampling. Patients have an indication for EBUS-TBNA.

Intervention: Patients will undergo an EBUS investigation followed by EUS-B in the same session. During this single scope procedure, lymph nodes that are suspected on prior CT-PET imaging and on subsequent ultrasound are sampled.

Main study endpoint: The main study parameter is the sensitivity for locoregional disease (N2, N3, T4 disease) of complete endosonographic staging (by EBUS-TBNA and EUS-B-FNA) in comparison with EBUS staging alone.

ELIGIBILITY:
Inclusion Criteria:

* (Suspected) NSCLC;
* Indication for mediastinal nodal assessment;
* Suspected mediastinal lymph nodes within reach of EBUS;
* Age 18 years or older;
* Clinically fit to undergo surgical resection of the lung tumor;
* Provision of a written informed consent;

Exclusion Criteria:

* Mediastinal re-staging after neo-adjuvant treatment;
* Indication for EUS other than mediastinal staging, eg a for malignancy
* suspected left adrenal;
* Active malignancy with a life expectancy of less than two years;
* Former therapy for lung cancer (chemotherapy, radiotherapy or surgery);
* Technical contraindication for EBUS or EUS (eg, esophagus stenosis);
* Pregnancy;
* Inability to consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with potentially operable and resectable NSCLC are eligible if there is an indication for mediastinal nodal sampling. Patients have an indication for EBUS-TBNA.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity for locoregional disease (N2, N3, T4 disease). | from inclusion untill either pathological proof of mediastinal metastases by endospnography or 1 week after surgical verification
  Sensitivity is defined as number of true positives (pathologic proof of a nodal metastases) divided by the number of true positives and false negatives (thoracotomy with nodal dissection is the reference standard to detect false negatives).
  The main study parameter is the sensitivity for locoregional disease (N2, N3, T4 disease) of complete endosonographic staging (by EBUS-TBNA and EUS-B-FNA) in comparison with EBUS staging alone.
  In the event of pathological proof of mediastinal metastases (N2/N3) by endosonography patients are classified as having locally advanced disease (stage III) and the study stops. When no mediastinal metastases are found by endosonography, surgical verification will take place (reference standard).

SECONDARY OUTCOMES:
Sensitivity for locally advanced disease (N2-3 metastases, T4). Systematic assessment and sampling of mediastinal lymph nodes versus PET-CT directed assessment of the mediastinum. | from inclusion untill either pathological proof of mediastinal metastases by endosonography or 1 week after surgical verification
  Sensitivity for locally advanced disease (N2-3 metastases, T4) of systematic assessment and sampling of mediastinal lymph nodes in comparison to PET-CT directed assessment of the mediastinum (ie targeted approach).

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (9):
- Belgium (2):
  - Onze-Lieve-Vrouwen-Ziekenhuis, Aalst
  - Universitair Ziekenhuis Leuven, Leuven
- Netherlands (7):
  - Academic Medical Center, Amsterdam, North Holland
  - Medisch Centrum Alkmaar, Alkmaar
  - Antoni van Leeuwenhoek ziekenhuis, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Universitair Medisch Centrum st Radboud, Nijmegen
  - Isala klinieken, Zwolle